CLINICAL TRIAL: NCT04878991
Title: Non-Selection Trial Comparing Metabolomics to Morphology Embryo Selection
Brief Title: Overture Metabolomics Non-Selection Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Overture Life (Industry)
Collaborators: New Hope Fertility Center (Other); Clinica Juana Crespo (Unknown)
Responsible Party: Principal Investigator, Dr. Jose Horcajadas, Principal Investigator, Overture Life
Other Study IDs: SUB-OVL-IRB-MTB-06.01.2021
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Infertility
Keywords: IVF; genetic screening; preimplantation genetic testing
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Treatment Group: Patients will undergo a routine IVF cycle. This will include ovarian stimulation, egg retrieval and fertilization of oocytes through intracytoplasmic sperm injection (ICSI). All fertilized oocytes will be cultured up to blastocyst for five to six days.
  Spent media will be collected on day 5-6 for all embryos reaching blastocyst on day 5, and on day 6 for those reaching blastocyst on day 6. The spent culture media will be sent to a lab for metabolomic analysis.
  For the embryo transfer, the best morphology blastocyst will be selected for transfer by the study embryologist. The embryo transfer outcome will be compared to the Metabolomics result to determine the NPV and PPV of Metabolomics vs implantation.
  Interventions: Diagnostic Test: Overture Metabolomics Embryo Selection

INTERVENTIONS:
Diagnostic Test: Overture Metabolomics Embryo Selection — Patients will have their embryos selected for transfer based on morphology alone. The embryo transfer outcome will be compared to the metabolomics result to determine the NPV and PPV of metabolomics vs implantation.

SUMMARY:
In this study, study investigators will collect embryo culture media on day 5 of vitro fertilization (IVF) culture, prior to vitrification and embryo transfer for testing via Metabolomic screening. Metabolomics is a new, non-invasive method of embryo selection which involves testing discarded embryo culture media for analytes secreted by the developing embryo. These analytes can be used to determine the implantation potential, and ploidy, of the embryo.

This study will take place at multiple locations in the United States and Spain.

DETAILED DESCRIPTION:
Patients will undergo ovarian stimulation, egg retrieval and fertilization of oocytes through intracytoplasmic sperm injection (ICSI). All fertilized oocytes will be cultured up to blastocyst for five to six days.

Spent media will be collected on day 5-6 for all embryos reaching blastocyst on day 5, and on day 6 for those reaching blastocyst on day 6. The spent culture media will be sent to a lab for metabolomic analysis. Details of sample collection and analysis are provided in Sections 6.3.1 & 6.3.2.

Single embryo transfer will be performed with the best morphology blastocyst being selected for transfer by the New Hope embryologist.

Approximately 8-11 days after the embryo transfer, the patient will return to the clinic for a serum pregnancy test. Should the test be negative, they will be closed out of the study. Should the test be positive, they will continue to be monitored.

The patient will return to the clinic at approximately 8 weeks after embryo transfer for a serum pregnancy test, and an ultrasound to detect fetal heartbeat. The outcome will be documented, and the patient monitored until 12 weeks of gestation at which time they will be closed from the study.

The embryo transfer outcome will be compared to MPI and MEI result to determine the NPV and PPV of metabolomics vs implantation.

ELIGIBILITY:
Inclusion Criteria:

* Women of any age, including egg donors. 50% will be <35 and the rest 35 and older.
* Signed Subject Consent Form. No inferior limit on number of eggs

Exclusion Criteria:

At the time of initial visit:

* Require or request PGT of any kind
* Low ovarian reserve defined as follicle stimulating hormone (FSH) >10 IU/L on day 2-4 of a prior menstrual cycle and anti-mullerian hormone (AMH) <15 pmol/L (or <2 ng/ml) within prior 12 months of cycle start

At the time of embryo selection:

-Patients without at least one embryo to transfer.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients recruited from an IVF center
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this non-selection study are negative predictive value (NPV) and positive predictive value (PPV) for MEI vs. PGT-A. | 8 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Jose Horcajadas, PhD, Principal Investigator — Overture Life; Santiago Munne, PhD, Principal Investigator — Overture Life
Locations (2):
- New Hope Fertility Center, New York, New York, United States
- Clinical Juana Crespo, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be presented at industry conferences, and published in peer reviewed journals.